CLINICAL TRIAL: NCT04861454
Title: Brassiere Brow Suture and Internal Browpexy as Disjunctive Upper Eyelid Blepharoplasty
Brief Title: Brassiere Brow Suture and Internal Browpexy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, Associate Professor, Benha University
Other Study IDs: Hamaky10
Record Dates: First submitted 2021-04-19; First posted 2021-04-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Eyelid Diseases
Keywords: blepharoplasty; browbexy
MeSH Terms: conditions — Eyelid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surgical: internal browbexy and brassier suture were done after blepharoplasty

SUMMARY:
Brow ptosis is a common problem. internal browbexy and brassier suture are common surgical approach

DETAILED DESCRIPTION:
upper eye transcutaneous blepharoplasty then combined browbexy and brassier suture are done

ELIGIBILITY:
Inclusion Criteria:

* brow ptosis and dermatochalasis

Exclusion Criteria:

* eyelid diseases and previous surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 18 years with dermatochalasis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
global aesthetic scale | 1 year
  calculate scale score from score 1 exceptional improvement to 5 worsening patient

CONTACTS AND LOCATIONS:
Overall Officials: tarek elhamaky, MD, Principal Investigator — Benha University
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates